CLINICAL TRIAL: NCT02512952
Title: Treatment of Periodontal Intrabony Defects Using Autologous Platelet Rich Fibrin and Titanium Platelet Rich Fibrin: A Randomized Clinical Comparative Study
Brief Title: Treatment of Periodontal Intrabony Defects Using Autologous Platelet Rich Fibrin vs Titanium Platelet Rich Fibrin
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Collaborators: The Oxford Dental College, Hospital and Research Center, Bangalore, India (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor and Head, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 224/2013-14
Record Dates: First submitted 2015-07-23; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Periodontitis
Keywords: Periodontal regeneration; Growth factors
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): SRP with Open flap debridement (OFD) alone for treating periodontal pocket
  Interventions: Procedure: Open flap debridement (OFD)
- Group 2 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF) placement into bone defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)
- Group 3 (Active Comparator): SRP with Open flap debridement (OFD) with Titanium Platelet rich fibrin (TPRF) placement into bone defect
  Interventions: Procedure: OFD with Titanium Platelet rich fibrin (TPRF)

INTERVENTIONS:
Procedure: Open flap debridement (OFD) — Oral prophylaxis followed by Open flap debridement (OFD)
  Arms: Group 1
Procedure: OFD with Platelet rich fibrin (PRF) — Oral prophylaxis followed by Open flap debridement (OFD) with Platelet rich fibrin (PRF) placement into the bone defect
  Arms: Group 2
Procedure: OFD with Titanium Platelet rich fibrin (TPRF) — Oral prophylaxis followed by Open flap debridement (OFD) with Titanium Platelet rich fibrin (TPRF) placement into the bone defect
  Arms: Group 3

SUMMARY:
Background: To compare the effectiveness of open flap debridement (OFD) alone and OFD along with either Autologous Platelet Rich Fibrin (PRF) or Titanium Platelet Rich Fibrin (TPRF) in the treatment of intrabony defects (IBDs).

Materials and methods: Study was conducted on subjects reporting to the Department of Periodontics, The Oxford Dental College and Hospital, Bangalore. 38 subjects with 90 periodontal IBDs of moderate to severe periodontitis were selected and assigned to OFD alone (group I) or OFD with Autologous PRF (group II) or OFD with TPRF (group III). In each subject, a minimum number of two sextants were present with probing pocket depths (PPD) ≥5mm in at least three teeth.

ELIGIBILITY:
Inclusion Criteria:

* presence of minimum 20 permanent teeth
* age group 20-55 years
* radiographic evidence of periodontal IBDs
* probing pocket depth (PPD) >5mm in minimum two sextants in at least three teeth
* clinical attachment (CA) loss of ≥ 3mm.

Exclusion Criteria:

* Systemically compromised subjects
* those on medications (corticosteroids/ bisphosphonate therapy) that may interfere with wound healing
* grade III tooth mobility
* smokers and alcoholic subjects
* pregnant and lactating mothers
* subjects who underwent periodontal treatment within a period of 1 year.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
defect depth reduction (DDR) | Change from baseline to 9 months
change in clinical attachment level (CAL) | Change from baseline to 9 months

SECONDARY OUTCOMES:
change in probing pocket depths (PPD) | Change from baseline to 9 months
change in plaque index (PI) | Change from baseline to 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Government Dental College and Research Institute, Bangalore, Karnataka
  - The Oxford Dental College, Bangalore, Karnataka